CLINICAL TRIAL: NCT01634204
Title: Is the Support of a Web-based Weight Loss Program Effective in Supporting Self-initiated Weight Loss and Lifestyle Changes?
Brief Title: Efficacy of a Web-based Weight Loss Program
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: KiloCoach e.U. (Other); University Hospital Regensburg (Other)
Responsible Party: Principal Investigator, Luzia Valentini, Dr. rer. nat., Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KiloCoach
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Overweight; Obese
Keywords: weight reduction; web-based intervention; cost-effective; overweight; obesity; cardiovascular risk
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KiloCoach (Experimental): Study subjects use the KiloCoach program on at least 4 days per week within the first half of the 6 months intervention period. In the second half, program usage is ad libitum.
  Interventions: Other: KiloCoach
- Control (No Intervention): Study subjects try to reduce body weight on their own, without participating in an organized weight loss program, over a period of 6 months.
  Interventions: Other: Control

INTERVENTIONS:
Other: KiloCoach — Study participants in this arm will use the program to record nutrition and physical activity on at least 4 days per week within the first and ad libitum within the second 3 months of the intervention period.
  Study visits will be conducted at baseline as well as after 1, 3 and 6 months. After 12 months a follow up visit will be conducted.
  Arms: KiloCoach
Other: Control — Study subjects try to reduce their body weight on their own. They are free to exercise and/or change nutritional habits. Not allowed is taking part in any structured weight loss program.
  Study visits will be conducted at baseline as well as after 1,3 and 6 months. A follow up visit will be conducted after 12 months.
  Arms: Control

SUMMARY:
Since overweight and obesity, a risk factor for various diseases, is a prevalent problem in the modern society, it is important to search for new strategies to counteract this. In contrast to in person support, the internet provides a low cost opportunity, which is able to reach a large part of the population. Therefore a web-based weight loss program may be an adequate mean for many people. Now it is hypothesised that a web-based weight loss program is able to support a reduction of body weight and weight-related cardiovascular risk factors effectively and to promote a healthier lifestyle. It is expected that program use, compared to a control group, results in greater reductions in body weight and cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* age 30-65 years
* body Mass Index: 27-39,9 kg/m2
* ECOG-Performance status degree 0 or 1
* basal internet skills
* private internet access
* signed informed consent

Exclusion Criteria:

* malign diseases
* major organ diseases
* inflammatory bowel diseases
* insulin - dependent diabetes mellitus
* pregnancy, breast feeding
* treatment of eating disorders (e.g. bulimia, anorexia nervosa) within past 5 years
* parallel participation in other weight loss programs or other trials
* weight loss > 5% within past 6 month
* chronic therapy with glucocorticoids
* subjects treated because of psychiatric disorders (e.g. schizophrenia, bipolar disorder) in the past
* subjects with expected non-compliance to protocol guidelines

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
body weight reduction in % | after 3 months

SECONDARY OUTCOMES:
body weight reduction in % | after 6 and 12 months
cardiovascular risk | after 3,6 and 12 months
  Cardiovascular risk is assessed by hsCRP, Fetuin A, LDL/HDL-ratio, waist-to-hip-ratio, HOMA-IR, blood pressure, body mass index, lean body mass (LBM), fat mass (FM), body cell mass (BCM.)
Quality of life | after 3,6 and 12 months
  Quality of life is assessed by "Obesity and Weight-Loss Quality of Life-Instrument" and "Weight related symptom measure".
Nutrition and physical activity | after 3,6 and 12 months
  Nutritional intake (controls) is assessed by 3-day dietary protocols. Physical activity is assessed by "International physical activity questionnaire" (IPAQ-long), lower limb strength and phase angle.

CONTACTS AND LOCATIONS:
Overall Officials: Luzia Valentini, Doctor, Principal Investigator — Charite University, Berlin, Germany
Locations (3):
- KiloCoach e.U., Vienna, Austria
- Germany (2):
  - Charité- Universitätsmedizin Berlin, Berlin
  - University Hospital Regensburg, Regensburg

REFERENCES:
- [Background] Truby H, Baic S, deLooy A, Fox KR, Livingstone MB, Logan CM, Macdonald IA, Morgan LM, Taylor MA, Millward DJ. Randomised controlled trial of four commercial weight loss programmes in the UK: initial findings from the BBC "diet trials". BMJ. 2006 Jun 3;332(7553):1309-14. doi: 10.1136/bmj.38833.411204.80. Epub 2006 May 23. PMID 16720619
- [Background] Tate DF, Jackvony EH, Wing RR. A randomized trial comparing human e-mail counseling, computer-automated tailored counseling, and no counseling in an Internet weight loss program. Arch Intern Med. 2006 Aug 14-28;166(15):1620-5. doi: 10.1001/archinte.166.15.1620. PMID 16908795
- [Background] Harvey-Berino J, Pintauro S, Buzzell P, DiGiulio M, Casey Gold B, Moldovan C, Ramirez E. Does using the Internet facilitate the maintenance of weight loss? Int J Obes Relat Metab Disord. 2002 Sep;26(9):1254-60. doi: 10.1038/sj.ijo.0802051. PMID 12187404
- [Background] Harvey-Berino J, West D, Krukowski R, Prewitt E, VanBiervliet A, Ashikaga T, Skelly J. Internet delivered behavioral obesity treatment. Prev Med. 2010 Aug;51(2):123-8. doi: 10.1016/j.ypmed.2010.04.018. Epub 2010 May 15. PMID 20478333
- [Background] Tate DF, Wing RR, Winett RA. Using Internet technology to deliver a behavioral weight loss program. JAMA. 2001 Mar 7;285(9):1172-7. doi: 10.1001/jama.285.9.1172. PMID 11231746
- [Background] Krukowski RA, Harvey-Berino J, Ashikaga T, Thomas CS, Micco N. Internet-based weight control: the relationship between web features and weight loss. Telemed J E Health. 2008 Oct;14(8):775-82. doi: 10.1089/tmj.2007.0132. PMID 18954247
- [Background] Galanis DJ, Kolonel LN, Lee J, Le Marchand L. Anthropometric predictors of breast cancer incidence and survival in a multi-ethnic cohort of female residents of Hawaii, United States. Cancer Causes Control. 1998 Mar;9(2):217-24. doi: 10.1023/a:1008842613331. PMID 9578299
- [Background] Trentham-Dietz A, Newcomb PA, Egan KM, Titus-Ernstoff L, Baron JA, Storer BE, Stampfer M, Willett WC. Weight change and risk of postmenopausal breast cancer (United States). Cancer Causes Control. 2000 Jul;11(6):533-42. doi: 10.1023/a:1008961931534. PMID 10880035
- [Background] Goldstein DJ. Beneficial health effects of modest weight loss. Int J Obes Relat Metab Disord. 1992 Jun;16(6):397-415. PMID 1322866
- [Background] Longin R, Grasse M, Aspalter R, Waldherr K. Effectiveness of the online weight reduction program KiloCoach and comparison with other evaluated commercial direct intervention and online programs. Obes Facts. 2012;5(3):372-83. doi: 10.1159/000339726. Epub 2012 Jun 14. PMID 22722385